CLINICAL TRIAL: NCT00858312
Title: Role of Dairy Foods to Enhance Central Fat and Weight Loss With Moderate Energy Restriction in Overweight and Obesity Individuals
Brief Title: Dairy Foods and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FL49; DMI
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity
Keywords: dairy foods; weight loss; fat loss; metabolic regulation
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Diet with 3-4 servings of dairy-rich foods/day
  Interventions: Other: high dairy diet
- 2 (Placebo Comparator): Low Dairy < 1 serving of dairy food/day
  Interventions: Other: Low Dairy

INTERVENTIONS:
Other: high dairy diet — 12 week energy restriction with 3-4 servings of dairy foods/day.
  Arms: 1
Other: Low Dairy — less than 1 serving of dairy foods per day.
  Arms: 2

SUMMARY:
Obesity is a national epidemic with multiple causes and complex solutions. Research in both animals and humans has suggested that the inclusion of dairy foods into a moderate calorie restricted diet can increase weight loss and fat loss. Our proposed project extends these prior findings by determining, for the first time, how inclusion of dairy in a calorie-restricted diet changes the amount of visceral adiposity in overweight and obese subjects. The investigators also propose unique studies to evaluate the potential mechanism(s) by which dairy promotes weight and fat loss during dieting, through an examination of adipocyte size, gene expression, and inflammatory markers. The hypotheses under investigation are (1) that inclusion of dairy foods in a modest energy restricted diet will significantly increase body fat loss compared to a control diet; (2) that dairy products in a modest energy restricted diet will result in greater fat loss from intra-abdominal adipose tissue compared to the control, 3) components of dairy products up- or down-regulate the secretion of metabolically-relevant hormones during the postprandial and inter-meal periods, 4) dairy products will promote satiety and/or satiation, 5) dairy foods reduce adipocyte differentiation and/or enhance adipocyte apoptosis, leading to concomitant white adipose tissue (WAT) expression changes for genes playing a role in these processes, 6) dairy foods will reduce adipocyte lipid storage and enhance pathways associated with thermogenesis and mitochondrial function in WAT, as reflected in gene expression changes and reduced adipocyte size, and 7) dairy foods included in a modest energy restricted diet will decrease inflammation in WAT and other tissues, thus decreasing circulating cytokines, increasing zinc status, decreasing expression of inflammatory markers in WAT, and reducing WAT macrophage infiltration.

DETAILED DESCRIPTION:
84 overweight and overweight and obese adult males and females will be recruited from the faculty, staff, and student populations at University of California-Davis as well as the greater Davis and Sacramento communities. Each intervention arm will require 42 adults; 35 for statistical power on weight loss + 14 more for attrition during the weight loss intervention. Statistical power for fat loss requires only 20 subjects/treatment arm. Subjects will be enrolled in 7 cohorts of 12 each and will be randomly assigned to either control or dairy diets. Subjects will meet the following additional inclusion and exclusion criteria:

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 28 -3 4.9 kg/m2
* Age 20-45 years for females, age 20-50 for males
* Low calcium diet (determined by food frequency and diet history): < 1 serving of dairy foods and total dietary Ca intake from all sources not to exceed 600 mg/d .
* No more than 3 kg weight loss during past three months
* Negative pregnancy test at entry prior to DXA and abdominal CT scan; pregnancy testing will be repeated done at 6 weeks of diet intervention to insure that women do not become pregnant during the energy restriction period. Should a woman become pregnant she will be dismissed from the protocol. Pregnancy testing will also be done at the end of the study prior to DXA and abdominal CT scans

Exclusion Criteria:

* BMI<28or>37. BMI greater than 37 indicates another level of obesity and the potential for numerous obesity related endocrine changes and substrate utilization abnormalities.

  * Type II diabetes requiring the use of any oral anti-diabetic agent and/or insulin (because of confounding effects on body weight regulation).
  * Fasting glucose > 110 mg/dl.
  * Adverse response to study foods (lactose intolerance, dairy intolerance, dairy allergy; this will be determined by self-report.
  * High calcium diet (determined by food frequency and diet history): Greater than 600 mg calcium per day from all sources (Ca supplements, dairy foods and other dietary sources).
  * History or presence of significant metabolic disease which could impact on the results of the study (i.e. endocrine, hepatic, renal disease).
  * Use of hypertension or lipid altering medications.
  * Resting blood pressure > 160/100 mg/Hg
  * Total cholesterol > 300mg/dl or triglyceride value > 400 mg/dl or LDL > 160 mg/dl.
  * History of eating disorder
  * Presence of active gastrointestinal disorders such as malabsorption syndromes
  * Pregnancy or lactation
  * Use of obesity pharmacotherapeutic agents within the last 12 weeks
  * Use of over-the-counter anti-obesity agents (e.g. those containing phenylpropanolamine, ephedrine and/or caffeine) within the last 12 weeks
  * Use of calcium supplements in the past 12 weeks
  * Recent (past four weeks) initiation of an exercise program
  * Recent (past twelve weeks) initiation of hormonal birth control or change in hormonal birth control regimen
  * Use of tobacco products.
  * Exercise more than 30 minutes/day - greater than this may influence substrate utilization.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in body weight | measured at end of run-in diet and after 12 weeks of study diet
  Weight measured in kg
Change in body fat | measured at end of run-in diet and after 12 weeks of study diet
  Total body fat assessed using dual energy X-ray absorptiometry (DXA)
Change in intra-abdominal adipose tissue (IAAT) | measured at end of run-in diet and after 12 weeks of study diet
  Intra-abdominal adipose tissue IAAT volume measured in cubic centimeters using computed tomography (CT) transabdominal slices

SECONDARY OUTCOMES:
Change in subcutaneous adipose cell number and size | measured at end of run-in diet and after 12 weeks of study diet
  Subcutaneous adipose tissue samples obtained by needle biopsy prepared for histological examination of cell number and size in square micrometers (uM2)
Change in subcutaneous adipose tissue inflammation | measured at end of run-in diet and after 12 weeks of study diet
  Subcutaneous adipose tissue samples obtained by needle biopsy were prepared for histological examination of the number of macrophages.
Change in subcutaneous adipose tissue gene expression | measured at end of run-in diet and after 12 weeks of study diet
  Subcutaneous adipose tissue samples obtained by needle biopsy were prepared for RNA extraction
Change in insulin | measured at end of run-in diet and after 12 weeks of study diet
  Serum insulin concentration (pmol/L) measured using multiplex technology.
Change in glucose | measured at end of run-in diet and after 12 weeks of study diet
  Plasma glucose concentration (mmol/L) measured using standard clinical methods
Change in total cholesterol | measured at end of run-in diet and after 12 weeks of study diet
  Serum cholesterol concentration (mmol/L) measured using standard clinical methods
Change in low density lipoprotein (LDL) cholesterol | measured at end of run-in diet and after 12 weeks of study diet
  Serum LDL cholesterol concentration (mmol/L) measured using standard clinical methods
Change in high density lipoprotein (HDL) cholesterol | measured at end of run-in diet and after 12 weeks of study diet
  Serum HDL cholesterol concentration (mmol/L) measured using standard clinical methods
Change in vitamin D (calciferol) metabolites | measured at end of run-in diet and after 12 weeks of study diet
  Serum 25-OH Vitamin D (nmol/L) and 1,25 (OH)2 vitamin D concentration (pmol/L) measured using radioimmunoassay (RIA)
Change in leptin | measured at end of run-in diet and after 12 weeks of study diet
  Serum leptin concentration (ng/ml) measured using multiplex technology.
Change in adiponectin | measured at end of run-in diet and after 12 weeks of study diet
  Serum adiponectin concentration (ug/mL) measured using multiplex technology.
Change in inflammatory cytokines | measured at end of run-in diet and after 12 weeks of study diet
  Serum inflammatory cytokine concentration (pg/mL) measured using multiplex technology.
Change in high sensitivity C-reactive protein (hs-CRP) | measured at end of run-in diet and after 12 weeks of study diet
  Serum hs-CRP concentration (mg/L) measured using immunoassay
Change in amylin | measured at end of run-in diet and after 12 weeks of study diet
  Serum amylin concentration measured using multiplex technology.
Change in peptide-YY (PYY) | measured at end of run-in diet and after 12 weeks of study diet
  Serum PYY concentration measured using multiplex technology.
Change in cholecystokinin (CCK) | measured at end of run-in diet and after 12 weeks of study diet
  Serum CCK concentration measured using radioimmunoassay
Change in glucagon like peptide-1 (GLP-1) | measured at end of run-in diet and after 12 weeks of study diet
  Serum GLP-1 concentration measured using multiplex technology.
Change in gastric inhibitory peptide (GIP) | measured at end of run-in diet and after 12 weeks of study diet
  Serum GIP concentration measured using multiplex technology.
Change in sun exposure | measured twice per week for 12 consecutive weeks of study diet
  Sun exposure was estimated from a personal diary kept weekly for recording time outdoors in hourly increments from 7 am to 7 pm combined with a clothing and sunscreen use standard key. Ultraviolet B (UVB) data was collected from various regional climate stations enrolled in the USDA UVB Monitoring Research Program (UVMRP).
Change in skin reflectance | measured at end of run-in diet and after 12 weeks of study diet
  Spectrophotometric measure of skin pigmentation for assessment of vitamin D status
Change in salivary cortisol in response to a meal | 15 minutes before, and 30, 45 and 60 min after lunch
  Cortisol concentration measure by high sensitivity enzyme linked immunoassay (nmol/L)
Change in salivary cortisol in response to a buffet | before and 30 min after buffet
  Cortisol concentration measure by high sensitivity enzyme linked immunoassay (nmol/L)
Change in salivary cortisol in response to weight loss | measured at end of run-in diet and after 12 weeks of study diet
  Cortisol concentration measure by high sensitivity enzyme linked immunoassay (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Marta D Van Loan, Ph.D., Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Van Loan MD, Keim NL, Adams SH, Souza E, Woodhouse LR, Thomas A, Witbracht M, Gertz ER, Piccolo B, Bremer AA, Spurlock M. Dairy Foods in a Moderate Energy Restricted Diet Do Not Enhance Central Fat, Weight, and Intra-Abdominal Adipose Tissue Losses nor Reduce Adipocyte Size or Inflammatory Markers in Overweight and Obese Adults: A Controlled Feeding Study. J Obes. 2011;2011:989657. doi: 10.1155/2011/989657. Epub 2011 Sep 14. PMID 21941636
- [Background] Witbracht MG, Laugero KD, Van Loan MD, Adams SH, Keim NL. Performance on the Iowa Gambling Task is related to magnitude of weight loss and salivary cortisol in a diet-induced weight loss intervention in overweight women. Physiol Behav. 2012 May 15;106(2):291-7. doi: 10.1016/j.physbeh.2011.04.035. Epub 2011 Apr 30. PMID 21565212
- [Background] Witbracht MG, Van Loan M, Adams SH, Keim NL, Laugero KD. Dairy food consumption and meal-induced cortisol response interacted to influence weight loss in overweight women undergoing a 12-week, meal-controlled, weight loss intervention. J Nutr. 2013 Jan;143(1):46-52. doi: 10.3945/jn.112.166355. Epub 2012 Nov 28. PMID 23190756
- [Background] Piccolo BD, Dolnikowski G, Seyoum E, Thomas AP, Gertz ER, Souza EC, Woodhouse LR, Newman JW, Keim NL, Adams SH, Van Loan MD. Association between subcutaneous white adipose tissue and serum 25-hydroxyvitamin D in overweight and obese adults. Nutrients. 2013 Aug 26;5(9):3352-66. doi: 10.3390/nu5093352. PMID 24067385
- [Background] Piccolo BD, Keim NL, Fiehn O, Adams SH, Van Loan MD, Newman JW. Habitual physical activity and plasma metabolomic patterns distinguish individuals with low vs. high weight loss during controlled energy restriction. J Nutr. 2015 Apr;145(4):681-90. doi: 10.3945/jn.114.201574. Epub 2015 Jan 28. PMID 25833772
- [Derived] Krishnan S, Adams SH, Witbracht MG, Woodhouse LR, Piccolo BD, Thomas AP, Souza EC, Horn WF, Gertz ER, Van Loan MD, Keim NL. Weight Loss, but Not Dairy Composition of Diet, Moderately Affects Satiety and Postprandial Gut Hormone Patterns in Adults. J Nutr. 2021 Jan 4;151(1):245-254. doi: 10.1093/jn/nxaa327. PMID 33245130
- [Derived] Piccolo BD, Hall LM, Stephensen CB, Gertz ER, Van Loan MD. Circulating 25-Hydroxyvitamin D Concentrations in Overweight and Obese Adults Are Explained by Sun Exposure, Skin Reflectance, and Body Composition. Curr Dev Nutr. 2019 May 27;3(7):nzz065. doi: 10.1093/cdn/nzz065. eCollection 2019 Jul. PMID 31304455